CLINICAL TRIAL: NCT04965961
Title: Plasma and Exosome Proteomic Changes Associated With Augmented Erythropoiesis and Muscle Contractions.
Brief Title: The Effect of Micro-doses Erytropoietin on Exercise Capacity in Male and Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Nikolai Nordsborg, Professor, Head of Department, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-18013069
Record Dates: First submitted 2021-06-28; First posted 2021-07-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sports Drug Abuse
Keywords: erythropoeitin; doping

STUDY DESIGN:
Intervention Model Description: Explorative
Who Masked: Participant, Investigator
Masking Description: An algorithm was created using randomizer.org
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant human erythropoietin treatment (Experimental): Participants receive intravenous injections of 9 International Units per kg bodyweight epoetin-β (NeoRecormon, Roche, Mannheim, Germany) three times per week for four weeks on non-consecutive days. Subjects receive tablets with 80mg iron (Tardyferon, Pierre Fabre Pharme GmbH, Freiburg, Germany) to ensure sufficient iron stores for the expected increase in erythropoeisis.
  Interventions: Drug: EPO
- Control group (Placebo Comparator): Participants receive intravenous injections of ~0,5 mL saline (NaCl 0,9%) three times per week for four weeks on non-consecutive days.
  Interventions: Other: Control group - saline injection

INTERVENTIONS:
Drug: EPO — Please refer to the arm description
  Arms: Recombinant human erythropoietin treatment
Other: Control group - saline injection — Please refer to the arm description
  Arms: Control group

SUMMARY:
Recombinant human erythropoietin (rHuEPO) regimen enhances maximal oxygen consumption (VO2max), but the effect of micro-doses on maximal and submaximal performance is not clear and detection of micro-doses is difficult with current methods. This study investigated whether micro-doses of rHuEPO enhances maximal and endurance performance in males and females.

DETAILED DESCRIPTION:
In a randomized, double-blind, placebo-controlled design, 48 trained adults (24 females, 24 males) receive either recombinant human erythropoietin (rHuEPO; epoetin-β, 9 IU/kg, n = 24, (12 females, 12 males)) or placebo (0,9% NaCl, n = 24, (12 females, 12 males)) three times per week for four weeks. Before the intervention, time trial performance and maximal oxygen uptake will be assessed. Three and five days after the last injection, time trial performance and maximal oxygen uptake will be determined to assess the effect of the rHuEPO administration. In addition, total hemoglobin mass and intravascular volumes will be determined via the carbon monoxide rebreathing method in duplicate measures.

ELIGIBILITY:
Inclusion Criteria:

* Relative maximum oxygen uptake (VO2-max) of at least 50 ml O2/min/kg for male participants and 45 ml O2/min/kg for female participants

Exclusion Criteria:

* Age
* Insufficient fitness level
* Blood donation 3 months prior to enrollment
* Altitude exposure 2 months before enrollment
* Hypertension

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in maximal oxygen uptake | Change from baseline to 5 days after last injection
  Change from baseline maximal aerobic capacity 5 days after last injection. Measured via an exhaustive incremental cycle ergometer test.
Change in time trial performance | Change from baseline to 3 days after last injection
  Change from baseline endurance exercise performance 3 days after last injection. Measured via a preloaded 400 kcal time-trial.
Change in total hemoglobin mass | Change from baseline to 3 days after last injection
  Change from baseline total hemoglobin mass 3 days after last injection. Measured by the carbon monoxide rebreathing method.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Fully anonymous data can be shared with other researchers.

REFERENCES:
- [Derived] Breenfeldt Andersen A, Bejder J, Bonne TC, Graae J, Seier S, Nordsborg NB. Changes in Immature Reticulocytes Aid the Indirect Detection of Microdose Recombinant Erythropoietin Use in Men and Women. Med Sci Sports Exerc. 2023 Sep 1;55(9):1695-1705. doi: 10.1249/MSS.0000000000003197. Epub 2023 Apr 24. PMID 37095637
- [Derived] Breenfeldt Andersen A, Graae J, Bejder J, Bonne TC, Seier S, Debertin M, Eibye K, Hostrup M, Nordsborg NB. Microdoses of Recombinant Human Erythropoietin Enhance Time Trial Performance in Trained Males and Females. Med Sci Sports Exerc. 2023 Feb 1;55(2):311-321. doi: 10.1249/MSS.0000000000003052. Epub 2022 Nov 1. PMID 36317927